CLINICAL TRIAL: NCT04193033
Title: Evaluation of Implementing FLOW: Transitioning Stabilized Mental Health Patients to Management in Primary Care (PEC 19-302)
Brief Title: Evaluation of Implementing FLOW
Acronym: FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PEX 19-004
Record Dates: First submitted 2019-11-25; First posted 2019-12-10 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Mental Health
Keywords: mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomization will be at the site level. All 9 sites will receive the intervention, using a stepped wedge design. Sites will be randomly allocated to one of three cohorts, and all sites within a cohort will receive the intervention at the same time. Cohort start dates will be offset by three months to allow examination of time effects.
Masking Description: Because this is a stepped wedge design QI clinical trial, masking is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FLOW intervention (Experimental): Sites receive the FLOW program, including internal and external facilitation, use of the FLOW online report to identify patients, patient and provider education materials, a medical record template, and regular data tracking and feedback about the process.
  Interventions: Other: FLOW intervention
- Waitlist until Time 2 (No Intervention): Arm 2: In this stepped wedge design, sites will be randomized to receive the FLOW intervention at Time 1, or to be in a waitlist until Time 2.
- Waitlist until Time 3 (No Intervention): Arm 3: In this stepped wedge design, sites will be randomized to receive the FLOW intervention at Time 1, or to be in a waitlist until Time 3.

INTERVENTIONS:
Other: FLOW intervention — The FLOW program, including internal and external facilitation, use of the FLOW online report to identify patients, patient and provider education materials, a medical record template, and regular data tracking and feedback about the process.
  Arms: FLOW intervention

SUMMARY:
Adequate access to mental health is one of the most important problems facing the VA and VISN 19. Mental health patients who are stabilized and recovered should be transitioned back to primary care to increase availability in mental health for new patients, and to signal to recovered patients that they are successfully recovered. Because there are currently no methods to identify who is recovered or tools and processes to assist in transitions, few patients 'graduate' mental health. The FLOW program consists of an algorithm to identify patients who are potentially appropriate for transition, a user-friendly online report to communicate this information to providers, materials to explain this process to patients and providers, and an electronic medical record (EMR) note template to document the transition. The investigators are partnering with VISN 19 to evaluate this program using a stepped wedge design with 9 sites randomly allocated into 3 steps in the wedge. Sites will receive an evidence-based implementation facilitation approach. The investigators will evaluate the number of patients transitioned, success of those transitions, and patient and provider satisfaction.

DETAILED DESCRIPTION:
Our study sites requested that we pause implementation due to clinical efforts and site disruption related to COVID-19. Date of study resumption is unclear.

Adequate access to mental health is one of the most important problems facing the VA and VISN 19. Mental health patients who are stabilized and recovered should be transitioned back to primary care to increase availability in mental health for new patients, and to signal to recovered patients that they are successfully recovered. Because there are currently no methods to identify who is recovered or tools and processes to assist in transitions, few patients 'graduate' mental health. The FLOW program consists of an algorithm to identify patients who are potentially appropriate for transition, a user-friendly online report to communicate this information to providers, materials to explain this process to patients and providers, and an electronic medical record (EMR) note template to document the transition. The investigators are partnering with VISN 19 to evaluate this program using a stepped wedge design with 9 sites randomly allocated into 3 steps in the wedge. Sites will receive an evidence-based implementation facilitation approach. The investigators will evaluate the number of patients transitioned, success of those transitions, and patient and provider satisfaction.

Specific aims for this proposal are:

1. To evaluate the impact of FLOW, using the evaluation framework RE-AIM, including:

   1. Reach of the program: % of clinic patients transitioned to PC using FLOW
   2. Effectiveness: successful transition to primary care and impact on clinic access for future patients
   3. Adoption: percent of providers in the selected clinics transitioning patients to primary care
   4. Implementation: use of all FLOW components
   5. Maintenance: sustainment of FLOW after withdrawal of external facilitation
2. To evaluate structural and process implementation factors, including organizational readiness to change, staffing levels, interservice agreements about care, leadership support, and internal facilitation.

ELIGIBILITY:
Inclusion Criteria:

* This study uses site-level randomization
* Sites must be VA sites with substantial numbers of mental health patients

  * VA medical centers or large or very large community based outpatient clinics

Exclusion Criteria:

* Non-VA sites and CBOCs smaller than large

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie E Hundt, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This QI project uses site-level randomization and a stepped wedge design. Individual participants are not recruited into the study and do not provide informed consent. The quality improvement intervention is rolled out across sites, and the primary outcomes include access to care, which data are freely available to all VA investigators via the VA administrative and clinical databases.

REFERENCES:
- [Derived] Hundt NE, Kim B, Plasencia M, Amspoker AB, Walder A, Yusuf Z, Nagamoto H, Tsao CG, Smith TL. Factors associated with successful FLOW implementation to improve mental health access: a mixed-methods study. Transl Behav Med. 2024 Nov 25;14(12):693-702. doi: 10.1093/tbm/ibae050. PMID 39326034
- [Derived] Smith TL, Yusuf ZI, Kim B, Amspoker AB, Hundt NE. An external facilitation case study analysis of an implementation trial of FLOW: A program for improving the transition of patients with mental health disorders back to primary care. Psychol Serv. 2024 Aug 22. doi: 10.1037/ser0000898. Online ahead of print. PMID 39172402

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sites
Groups:
- FLOW Intervention: Sequence 1: 12 months of FLOW implementation, then 12 months of maintenance.
  Sites received the FLOW program, including internal and external facilitation, use of the FLOW online report to identify patients, patient and provider education materials, a medical record template, and regular data tracking and feedback about the process. Because this is a site-level trial, participants and providers were not directly enrolled in the trial.
  FLOW intervention: The FLOW program, including internal and external facilitation, use of the FLOW online report to identify patients, patient and provider education materials, a medical record template, and regular data tracking and feedback about the process.
- Waitlist Until Time 2: Sequence 2: 3 months of usual care, 12 months of FLOW implementation, then 9 months of maintenance
- Waitlist Until Time 3: Sequence 3: 6 months of usual care, 12 months of FLOW implementation, then 6 months of maintenance
Period: Overall Study
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Started | NA; 3 sites (Data only collected at site level - not participant level) | NA; 3 sites (Data only collected at site level - not participant level) | NA; 3 sites (Data only collected at site level - not participant level)
Completed | NA; 3 sites (Data only collected at site level - not participant level) | NA; 3 sites (Data only collected at site level - not participant level) | NA; 3 sites (Data only collected at site level - not participant level)
Not Completed | NA; 0 sites | NA; 0 sites | NA; 0 sites

BASELINE CHARACTERISTICS:
Population: This data was not collected for site level assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: Sites] — Population: Data only collected at site level, not participant level.

OUTCOME MEASURES:

1. Primary Outcome: Reach: Percent of Specialty Mental Health Patients Transitioned to Primary Care
Description: Percent of mental health patients in each of the participating clinics who are transitioned to primary care through use of the FLOW intervention, based upon electronic medical record data documenting this transition
Time Frame: Change from baseline to 12 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Percent of mental health patients
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Percent of mental health patients | 1.41 (.82) | .77 (.62) | 1.89 (1.56)
Statistical Analysis 1: Comparison: FLOW Intervention vs Waitlist Until Time 2 vs Waitlist Until Time 3; Test type: Superiority; p = 0.001, Linear Growth Curve Model

2. Primary Outcome: Effectiveness of Intervention's Impact on Clinic Access
Description: Appointments freed up by FLOW consistent discharges from mental health clinics, by site
Time Frame: Change from baseline to 12 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Appointment slots
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Appointment slots | 148.7 (98.69) | 222.33 (337.32) | 354.2 (242.49)
Statistical Analysis 1: Comparison: FLOW Intervention vs Waitlist Until Time 2 vs Waitlist Until Time 3; Test type: Superiority; p = 0.012, t-test, 2 sided

3. Primary Outcome: Adoption: Percent of Mental Health Providers Who Use FLOW Intervention
Description: Percent of mental health providers who use the FLOW intervention for at least 3 patients, compared to the total number of mental health providers in the participating clinics
Time Frame: 12 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Percent of providers
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Percent of providers | 14.24 (12.98) | 8.09 (7.33) | 8.47 (4.24)
Statistical Analysis 1: Comparison: FLOW Intervention vs Waitlist Until Time 2 vs Waitlist Until Time 3; Test type: Superiority; p = 0.66, ANOVA

4. Primary Outcome: Implementation Fidelity to the Protocol
Description: Percent of all FLOW components implemented as designed, based upon the items in the FLOW implementation checklist
Time Frame: 12 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Percent of FLOW components
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Percent of FLOW components | 100 (0) | 100 (0) | 100 (0)

5. Secondary Outcome: Maintenance of Effectiveness of Intervention's Impact on Clinic Access
Description: Encounter slots 'freed up' by FLOW discharges
Time Frame: 12-18 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Appointment slots
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Appointment slots | 171.73 (50.67) | 81.26 (95.76) | 147 (140.36)
Statistical Analysis 1: Comparison: FLOW Intervention vs Waitlist Until Time 2 vs Waitlist Until Time 3; Test type: Superiority; p = .49, Linear Growth Curve Model; Time was included as a fixed effect and both time and intercept were included as random effects

6. Secondary Outcome: Maintenance of Implementation Fidelity to the Protocol
Description: Percent of all FLOW components implemented as designed, based upon the items in the FLOW implementation checklist, from 12 to 24 months
Time Frame: 12-24 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Percent of FLOW components
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Percent of FLOW components | 100 (0) | 100 (0) | 100 (0)

7. Secondary Outcome: Maintenance of Reach: Percentage of Specialty Mental Health Patients Transitioned to Primary Care
Description: Percent of mental health patients in each of the participating clinics who are transitioned to primary care through use of the FLOW intervention, based upon electronic medical record data documenting this transition, during the maintenance period
Time Frame: from 12-24 months
Population: Data only collected at site level - not participant level
Measure: Mean (Standard Deviation); unit: Percent of mental health patients
Units Other Than Participants: Sites
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Sites) | 3 | 3 | 3
Percent of mental health patients | 2.95 (2.13) | 1.08 (1.25) | 2.59 (2.13)
Statistical Analysis 1: Comparison: FLOW Intervention vs Waitlist Until Time 2 vs Waitlist Until Time 3; Test type: Superiority; p = 0.06, t-test, 2 sided — Paired t-test, alpha = .05

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored.
Description: Adverse Events were not collected in this site-level randomized trial. This implementation project sought to influence provider behavior; patients were not directly enrolled.
Arm/Group | FLOW Intervention | Waitlist Until Time 2 | Waitlist Until Time 3
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Because this was a cluster randomized stepped wedge trial in which 9 sites were randomized to receive the intervention at different times, we have no comparison sites which never received the intervention and the overall sample size (n = 9) was small. Additionally, the 9 sites were all in one VA Veterans Integrated Service Network (VISN), under the same VISN leadership, so some informal spread of information about the intervention via informal networks may have occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04193033/Prot_SAP_000.pdf